CLINICAL TRIAL: NCT00536393
Title: Phase III Study of Treatment of Disseminated and Agressive Lymphoma R CHOP Versus R CLOP( With Liposomal Doxorubicin)
Brief Title: Treatment of Disseminated High Grade Lymphoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOELAMS 0804
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-09

CONDITIONS: Lymphoma
Keywords: diffuse larg cells lymphoma; chemotherapy; toxicity; diffuse high grade lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxorubicine (Active Comparator): CHOP 8 courses every 21 days
  Interventions: Drug: Doxorubicin
- Doxorubicine pegylated (Experimental): CLOP 8 courses every 21 days
  Interventions: Drug: Doxorubicin pegylated

INTERVENTIONS:
Drug: Doxorubicin
  Arms: Doxorubicine
Drug: Doxorubicin pegylated
  Arms: Doxorubicine pegylated

SUMMARY:
Interest of the use of pegylated liposomal doxorubicin (caélyx)

DETAILED DESCRIPTION:
R CHOP is a good standard in the treatment of diffuse high grade lymphoma. Howeverin elderly patients it is often toxic, specially with haematologic and cardiac toxicities.

ELIGIBILITY:
Inclusion Criteria:

* high grade lymphoma
* disseminated
* > 60 years old and < 75
* informed consent signed
* cardiac state compatible with antracyclin
* ECOG </= 2

Exclusion Criteria:

* patients > 75 years old
* Cardiac insufficiency

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2000-10; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
hematologic toxicity | 6 months

SECONDARY OUTCOMES:
response rate | 6 months
EFS and OS | 6 months
Cardiac toxicity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CARTRON, Dr, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Clinique Victor Hugo, Le Mans, France